CLINICAL TRIAL: NCT04767425
Title: Implementation of Image Guided Brachytherapy in Treatment of Patients With Locally Advanced Cancer Cervix
Brief Title: Image Guided Brachytherapy in Locally Advanced Cancer Cervix
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fatma Ahmed Abdelfatah Rikabe (Other)
Collaborators: Sohag University (Other)
Responsible Party: Sponsor-Investigator, Fatma Ahmed Abdelfatah Rikabe, Assistant lecturer of clinical oncology, Sohag University
Organization: Sohag University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ٍSoh-Med-21-02-02
Record Dates: First submitted 2021-02-18; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Cancer Cervix
Keywords: cancer cervix , brachytherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Radiation: Brachytherapy

INTERVENTIONS:
Radiation: Brachytherapy — • 3D image-based cervical cancer brachytherapy will be delivered as 4 sessions x 7 Gy High Dose Rate (HDR) brachytherapy

SUMMARY:
This is non comparative prospective interventional study with some areas for observational research to implement based image guided adaptive cervical cancer brachytherapy ( BT ) combined with Intensity Modulated Radiotherapy ( IMRT ) / Volumetric Modulated Arc Therapy ( VMAT) external beam radiotherapy (EBRT) ± chemotherapy (ChT) , and to take advantage of its full potential.

DETAILED DESCRIPTION:
* Eligible patients will receive both external beam radiotherapy ( EBRT) and concomitant chemotherapy and brachytherapy ( BT). Summation of EBRT and BT doses will be performed by calculation of a biologically equivalent dose in 2 Gy per fraction (EQD2) using the linear-quadratic model with α/β = 10 Gy for tumor effects and α/β = 3 Gy for late normal tissue damage. The repair half time is assumed to be 1.5 hrs.
* EBRT will be delivered as IMRT/VMAT with daily cone beam Computed Tomography ( CT ) Image Guided Radiotherapy (IGRT) in 25 fractions with 1.8 Gy to a total dose of 45 Gy given in 5 weeks.
* 3D image-based cervical cancer brachytherapy will be delivered as 4 sessions x 7 Gy High Dose Rate (HDR) brachytherapy , with ''Pre-radiotherapy Magnetic Resonance Imaging ( MRI ) examination'' to provide sufficient information about tumor extent in three dimension (3D) at the time of diagnosis and ''BT MRI examination'' is alse needed to provide sufficient information about tumor/target extent at the time of brachytherapy with the applicators in place .

For EBRT ; Using the cumulative Dose-volume histograms ( DVH ) to ensure that minimum dose to the target 95%, maximum dose limited to 107%, also, the dose to the organ at risk will be kept to the minimum according to the Radiation therapy oncology group ( RTOG ) recommendation.

For BT ; Dose volume adaptation will be performed with the aim of dose escalation in large tumors (prescribed D90 > 85 Gy , Dose volume constraints (D2cc) were 70-75 Gy for rectum and sigmoid and 90 Gy for bladder.

Differential DVH, the dose standard deviations will be used to asses dose homogeneity.

The conformity index and dose gradient measure will be calculated . Collection of data : Data will be collected by doctor himself in Excel sheet . Statistics : numerical Data will be reported with mean , median , standard deviation & variance and represented with suitable graph like histograms and frequency polygon . Discrete data will be analyzed with suitable tests like Chi-square test & fisher's exact test and will represented with suitable graph like pie graph .

Inferential statistics will be reported with 95 confidence interval & A P-value <0.05 will be considered as statistically significant .

Survival analysis will be analyzed using the actuarial Kaplan Meier method , time will be calculated with date of diagnosis .

Data from patients who had not reached the endpoint at the time of last follow -up will be treated as censored observations

ELIGIBILITY:
Inclusion Criteria:

* • Pathological confirmation squamous carcinoma, adenocarcinoma or adeno-squamous carcinoma of the uterine cervix.

  * Locally advanced cervical cancer , Federation of Gynecology and Obstetrics staging system FIGO stage IB ,FIGO stage IIA , FIGO stage IIB , FIGO stage IIIA, FIGO stage and FIGO stage IVA (and nodal status according to TNM) in whom definitive radio-chemotherapy with curative intent is planned are qualified for the study .
  * No evidence of distant metastasis or other malignancy.
  * No other comorbid disease that would affect patient survival

Exclusion Criteria:

* • FIGO stage IA , FIGO stage and Distant metastatic disease or presence of other malignancy .

  * Presence of other comorbid disease that would affect patient survival

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — this study is gender based as it's aim is evaluation of image guided brachytherapy in management of cancer cervix which is disease limited to females .
Enrollment: 50 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Reduction of tumor size | "up to 3 months "
  Complete response , defined as the disappearance of all evidence of disease by physical examination and MRI pelvis

SECONDARY OUTCOMES:
survival rates | " 2 years "
  survival rates including disease free survival, overall survival
Degree of toxicity | "through study completion, an average of 2 year"
  early and late treatment toxicity

IPD SHARING:
Plan to Share IPD: No